CLINICAL TRIAL: NCT01812863
Title: Pain Management in Children Undergoing Supracondylar Humerus Fracture Repair: Can a Local Supraclavicular Block Improve Their Postoperative Outcome?
Brief Title: Pain Management in Children Undergoing Supracondylar Humerus Fracture Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Our anesthesiologist was no longer available to assist.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-14957
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-01

CONDITIONS: Humeral Fractures; Fractures, Closed
Keywords: Pain Management; Child; Surgery
MeSH Terms: conditions — Humeral Fractures; Fractures, Closed; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supraclavicular Nerve Block (Experimental): Maximum dose of 5 mL of 0.25% bupivacaine, and we base the dose on a ml/ kg (0.2 ml/kg) with a maximum dose not to exceed 2.5 mg/kg. Bupivacaine is given with 1:200,000 epinephrine
  Interventions: Procedure: Supraclavicular nerve block
- No Nerve Block (Placebo Comparator): A band-aid will be placed on all patients where a supraclavicular nerve block would have been inserted, and parents will be asked to leave the band-aid on for 3 days to maintain the blindness to the treatment type by the patient.
  Interventions: Procedure: Supraclavicular nerve block

INTERVENTIONS:
Procedure: Supraclavicular nerve block — Following injection of morphine, an ultrasound-guided supraclavicular nerve catheter (Angiocath) will be placed in Group 2. All catheters will be placed by one of the anesthesiologist trained in regional pain control using a 25 mm linear US probe in a sterile fashion.
  If the examination is unchanged from preoperative assessment, an injection block using 5 ml of 0.25% bupivacaine with 1:200,000 epinephrine will be administered. Bupivacaine is a long acting local anesthetic that prevents nerve conduction and action potential initiation by decreasing the permeability of the neuronal membrane to sodium. We use a maximum dose of 5 mL of 0.25% bupivacaine, and we usually base the dose on a ml/kg (0.2 ml/kg) with a maximum dose not to exceed 2.5 mg/kg. This will be well below toxic levels.

SUMMARY:
The purpose of this study is to determine if US-guided supraclavicular anesthetic blocks reduce postoperative pain, use of rescue medication, and improve functional outcomes in children who underwent surgery for supracondylar humerus fractures.

DETAILED DESCRIPTION:
Forty six American Society of Anesthesiologists (ASA) class I or II patients between the ages of 2 and 10 years undergoing reduction of supracondylar humerus fractures will be enrolled in the study. From mid-May to the beginning of August, Lurie Children's (formerly Children's Memorial Hospital)historically has 50-70 supracondylar humerus fractures in children, and we expect an 80% recruitment rate for the study. A power analysis estimated that a sample size of 46 patients would have an 80% power at the 0.05 level of significance to detect a 50% reduction in the number of patients requiring rescue medication when comparing intravenous opioids and the ultrasound-guided supraclavicular nerve block (from approximately 80% to 40%).

After obtaining informed consent, the patients will be taken to the operating room where the procedure will be performed. Intraoperatively, patients will be randomly assigned to be in one of two groups. Randomization will be determined by block allocation with a 1:1 ratio with permuted, mixed blocks of 4 and 6 created randomly using a computer based randomization table. Randomization will be performed by one of the co-investigators. Preoperatively, patients will be assessed for neurovascular status by testing the patient's ability to make three movements: thumb extension (radial nerve), proximal interphalangeal joint (PIP) flexion (median nerve), and interossei function (ulnar nerve). Patients may be removed from the study after consent is given if removal of the cast prior to surgery reveals excessive swelling in the elbow, indicating an increased likelihood for development of compartment syndrome postoperatively. This determination will be made by the attending orthopaedic surgeon performing the procedure. Patients with an increased likelihood of developing compartment syndrome will be given narcotics to treat pain.

All patients will undergo a general anesthetic for the surgical procedure. Surgical anesthesia will be maintained using volatile anesthetics. Intraoperatively, while still under general anesthesia, Groups 1 and 2 will receive a standardized intravenous dose of 0.05 mg/kg of morphine in a total volume of 1 ml. Following injection of morphine, an ultrasound-guided supraclavicular nerve catheter (Angiocath) will be placed in Group 2. All catheters will be placed by one of the anesthesiologist trained in regional pain control using a 25 mm linear US probe in a sterile fashion.

Patients will be taken to the postoperative recovery room (PACU) area where they will be tested for nerve function after emergence from anesthesia. If the examination is unchanged from preoperative assessment, an injection block using 5 ml of 0.25% bupivacaine with 1:200,000 epinephrine will be administered. Bupivacaine is a long acting local anesthetic that prevents nerve conduction and action potential initiation by decreasing the permeability of the neuronal membrane to sodium. We use a maximum dose of 5 mL of 0.25% bupivacaine, and we usually base the dose on a ml/kg (0.2 ml/kg) with a maximum dose not to exceed 2.5 mg/kg. This will be well below toxic levels. A band-aid will be placed on all patients where a supraclavicular nerve block would have been inserted, and parents will be asked to leave the band-aid on for 3 days to maintain the blindness to the treatment type by the patient.

In the PACU, the patient will be evaluated for pain and discomfort by a member of the research team using the "Faces Pain Scale-Revised (FPS-R)" Other side effects such as nausea, vomiting, somnolence and respiratory depression will be noted. Any incidence of nausea and/or vomiting will be treated with 0.1 mg/kg (up to 4 mg) of ondansetron given intravenously.

The postoperative care unit staff is well versed in keeping children calm after anesthesia. There is a chance that the child may know which group they are in. However, due to the age of these children and the fact that they are just coming out of anesthesia, it is more likely that they will not understand what is happening and the implications of the interventions. It is also unlikely that it will affect the outcomes of requiring additional medication for pain in the PACU or at home. Likewise, it is unlikely that knowing the group would affect the range of motion outcome.

Families will be randomly contacted 7 times in the 36 hours approximately after the operation by nurses from the Collaborative Research Unit (CRU) to record a patient's pain score. Data will be analyzed using a time series analysis. Patients will be discharged with a standardized 5/325 mg dose of Norco to be taken every 4-6 hours. Patients are typically discharged the same day or after a brief overnight stay. Patients typically follow up in 1 week for a radiograph with the treating orthopaedic surgeon followed by pin removal at 3-4 weeks post-surgery. PT will begin if there is less than a 100 degree arc of motion at 6 weeks after pin removal and will involve ROM exercises per the PT discretion. A binary outcome will be recorded as to whether PT is necessary 6 weeks after the cast and pins are removed. Functional recovery will be measured 6 weeks after pin removal through ROM measurements. A pain score will also be taken at the follow-up visit 6 weeks after pin removal to measure long-term pain. Parents will be given a questionnaire before their child is discharged from the hospital. Part of the questionnaire is filled out while the child is still at the hospital. The rest of the questionnaire will be sent home with the parents to be filled out throughout the week following the operation. The contents of the questionnaire will be explained to the parents at the time that the questionnaire is handed out to ensure that they understand the questions. Parents will return the questionnaire at the 1 week follow up visit to give feedback data on any postoperative discomfort, any additional pain medications and also the overall satisfaction with the study design. All data obtained will be entered in an Excel® database. Statistical analysis will be carried out using the SPSS software® (Statistical Program for the Social Sciences), and a t-test will be performed with the data obtained. Primary outcome data will be the use of rescue medication in the immediate postoperative period. Secondary outcomes include pain scores, use of additional medication after leaving the hospital and range of motion at 9-10 weeks postoperatively. Analyzed data will include the duration of pain relief and retention of nerve functionality. We will also record and analyze the incidence of postoperative vomiting and respiratory distress in either group. We will carefully monitor and record for the development of compartment syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2 and 10 years old undergoing reduction and closed pinning of supracondylar humerus fractures
* Ability to obtain consent from the parents for participation in the study
* Patient has the ability to follow commands and train preoperatively the finger movements that are needed to determine nerve integrity.
* Written informed consent from the parent or guardian

Exclusion Criteria:

* Children with significant preoperative swelling in the elbow, as determined by the surgeon, that may lead to compartment syndrome
* Children with the potential for nerve entrapment as demonstrated by preoperative nerve deficit examination
* Children who have any contraindications (relative and absolute) to a supraclavicular block, including anticoagulation or coagulopathy, as well as patients that have active pulmonary disease that may exhibit respiratory compromise in response to potential phrenic nerve palsy or pneumothorax

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Rescue medication | In PACU following surgery
  We will record use of extra morphine in the PACU, if needed.

SECONDARY OUTCOMES:
Pain Scores | First 42 hours after surgery
  Patients have 8 pain scores recorded in the first 42 hours following surgery using the Faces Pain Scale-Revised (FPS-R)
Range of Motion | 9-10 weeks postoperatively
  Range of motion in the affected elbow will be measured 6 weeks after removal of pins
Physical therapy | 9-10 weeks postoperatively
  We will record whether patients need physical therapy for their elbow 6 weeks postoperatively
Vomiting | First 24 hours after surgery
  We record for vomiting in the PACU and in the first 24 hours post-op.

OTHER OUTCOMES:
Nausea | First 24 hours post-op
  We record for nausea in PACU and at home in the first 24 hours following surgery
Somnolence | First 24 hours post-op
  We record for somnolence in the PACU and in the first 24 hours post-op

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Janicki, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States